CLINICAL TRIAL: NCT02906722
Title: Efficacy of Nebulized Versus Intravenous Colimycin for Treating Ventilator-associated Pneumonia Caused by Gram-negative Multidrug-resistant Bacteria: a Prospective, Multicenter, Randomized and Double-blind Study
Brief Title: Nebulized and Intravenous Colistin in Ventilator Associated-pneumonia
Acronym: COLIVAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P130902; 2016-000389-41 (EudraCT Number)
Record Dates: First submitted 2016-08-12; First posted 2016-09-20 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2017-11

CONDITIONS: Ventilator-associated Pneumonia
Keywords: Nebulized colistin; Intravenous colistin; ventilator-associated pneumonia; multidrug resistance; Gram-negative bacteria
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients receive simultaneously nebulized colimycin every 8 h and intravenous placebo administered once, twice or 3 times per day according to renal function
  Interventions: Drug: Intravenous placebo; Drug: Nebulized colimycin
- Control group (Active Comparator): Patients receive simultaneously intravenous colimycin administered once, twice or 3 times per day according to function renal and nebulized placebo every 8 h
  Interventions: Drug: Intravenous colimycin; Drug: Nebulized placebo

INTERVENTIONS:
Drug: Intravenous colimycin — administration once, twice or 3 times per day according to renal function
  Arms: Control group
Drug: Intravenous placebo — administration once, twice or 3 times per day according to renal function
  Arms: Experimental group
Drug: Nebulized colimycin — Nebulization is performed with a vibrating plate nebulizer (Aeroneb® Solo) every 8h
  Arms: Experimental group
Drug: Nebulized placebo — Nebulization is performed with a vibrating plate nebulizer (Aeroneb® Solo) every 8h
  Arms: Control group

SUMMARY:
Few antimicrobials are available to treat ventilated associated pneumonia (VAP) caused by Gram negative multi-resistant (MDR) bacteria. Colimycin often remains the only active antibiotic. The aim of the study is to demonstrate the superiority of nebulized colimycin over intravenous colimycin to treat VAP caused by Gramnegative MDR bacteria.

DETAILED DESCRIPTION:
VAP is the most frequent nosocomial infection in critically ill patients and affects length of stay and cost in Intensive Care Unit. The increased incidence of nosocomial infections caused by MDR bacteria becomes a major health problem worldwide.

Nowadays, few antimicrobials are available to treat Gram negative MDR VAP. Colimycin often remains the only active antibiotic. Treating VAP by intravenous (IV) colimycin has two main limitations: risk of renal toxicity and low tissue penetration. Nebulization of colimycin offers the possibility of generating high lung tissue concentrations, rapid bactericidal effects and low systemic accumulation in experimental models. To date however, there is no study comparing clinical effectiveness of nebulized and intravenous colimycin.

We make the hypothesis that nebulized colimycin increases the clinical cure rate of VAP caused by Gram negative MDR bacteria compared to IV colimycin.

Primary Objective: To demonstrate the superiority of nebulized colimycin over intravenous colimycin for treating VAP caused by Gram-negative MDR bacteria.

Secondary Objectives:

1. To compare the microbiological cure rate at end of treatment
2. To compare the VAP recurrence rate after end of treatment
3. To compare the lung superinfection rate after end of treatment
4. To compare 28 day- and 90 day-mortality
5. To compare duration of mechanical ventilation
6. To compare length of ICU stay
7. To compare renal function during colimycin administration
8. To compare side effects resulting from colimycin nebulization and intravenous administration

Ancillary study:

In some centers, blood samples will be performed to measure colistin peak and trough plasma concentrations

Study design:

This is a randomized, multicenter, double-blind and phase III study

1. Randomization:

   Patients are randomly assigned to experimental group or control group:

   Control group: patients receive simultaneously intravenous colimycin and nebulized placebo.

   Experimental group: patients receive simultaneously nebulized colimycin and intravenous infusion of placebo.

   Dosing adjustment is according to renal function for intravenous infusion of colimycin or placebo.
2. Aerosol generation: Nebulization is performed with a vibrating plate nebulizer (Aeroneb® Solo) with following ventilator settings:

   * Constant flow and volume-controlled mode
   * Inspiratory/expiratory ratio of 1
   * Tidal volume of 6-8 ml/kg
   * Respiratory frequency of 12-18/min
   * End-inspiratory pause of 20% To standardize nebulization procedure, a checklist form is completed by the nurse in charge of the patient.
3. Duration of treatment:

   * 10 days in each group
   * In intubated patients, weaning test is authorized after 4 days of treatment. If patient is extubated, aerosols are discontinued whereas intravenous infusions are continued (placebo or antibiotic) until day 10
   * In tracheostomized patients: 10-day treatment for nebulized and intravenous therapy
4. Combined intravenous administration of other antimicrobials are authorized
5. Serum and microbiological samples

   * Serum creatinine measured daily from baseline to day 11
   * Lower respiratory tract specimens at day 5 and day 11 in intubated patients
6. Survival follow-up at day 28 and 90 days

Study population: Adult mechanical ventilated patients with VAP caused by Gram-negative MDR bacteria.

Sample size and Power consideration: Data will be analyzed with triangular test. Assuming a clinical cure rate at day 11 of 65% in the group treated with nebulized colimycin and of 45% in the group treated with intravenous colimycin, a mean sample size of 134 patients is required to provide 80% power, with a two-sided type I error rate of 5%. The 90th percentile of the number of patients to include is 196.

ELIGIBILITY:
Inclusion criteria

* Age older than 18 yr
* Invasive mechanical ventilation for more than 48 h Tracheostomized patients receiving intermittent mechanical ventilation can be included
* VAP caused by Gram-negative MDR bacteria resistant to all β-lactams and fluoroquinolones

Exclusion criteria

* Extrapulmonary Gram-negative MDR infection requiring intravenous colimycin
* VAP associated with bacteremia requiring combined treatment by nebulized and intravenous colimycin
* Hypersensitivity to colistimethate, colistin base, polymyxins and/or their excipients
* Porphyria
* Severe hypoxemia defined as PaO2 / FiO2< 100; if veno-venous ECMO is initiated, the patient can be included
* Severe brain injury (initial Glasgow coma score < 8) during the first 7 days before randomization
* Myasthenia
* cystic fibrosis
* Refusal to participate in the study
* Participation in any clinical study of a therapeutic investigational product within 30 days prior to the first day of inclusion
* No affiliation to social health insurance
* Patient under guardianship
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Clinical cure of VAP caused by Gram-negative multidrug resistant bacteria | At end of therapy visit (day11) or before day11 if treatment is considered as failed.
  Clinical cure is defined as:
  * resolution of clinical and biological signs of infection and improved radiological signs
  * and modified clinical pulmonary infection score (CPIS) less than 6
  * and negative culture of lower respiratory tract specimen or, successful weaning from invasive mechanical ventilation between day 5 and day 11
  * patient colonized with the same pathogen in the respiratory tract is considered as cured, if clinical and biological signs of infection resolved, radiological signs improved, CPIS < 6 and/or successful weaning from invasive mechanical ventilation has been obtained.

SECONDARY OUTCOMES:
Microbiological cure rate | At end of therapy visit (day11) or before day11 if treatment is considered as failed.
VAP recurrence rate | day 28
  VAP recurrence rate, defined as initial clinical cure of VAP with colimycin at day 11 followed by reappearance of clinical and biological signs of infection, CPIS greater than 6, and significant concentrations of Gram-negative MDR bacteria in lower respiratory tract specimen
Lung superinfection rate | day 11, day 28
  Lung superinfection rate defined as reappearance of VAP caused by pathogens other than Gram-negative MDR bacteria isolated from lower respi¬ratory tract specimens from day 11 to day 28
Mortality | day 28 and day 90
Duration of mechanical ventilation | Participants will be followed for the duration of ICU stay, an expected average of 3 weeks
Length of ICU stay | Participants will be followed for the duration of ICU stay, an expected average of 2 months
Renal function during colimycin administration | from Day 1 to Day 11
  Renal function is assessed by measuring daily serum creatinine during treatment period. Colimycin-induced renal function impairment is defined as an increase in serum creatinine level more than 1.5 times the pretreatment value
Side effects resulting from colimycin nebulization | from Day 1 to Day 11
Side effects resulting from colimycin intravenous administration | from Day 1 to day 28

OTHER OUTCOMES:
Colistin plasma concentrations | from Day 3 and Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Qin LU, MD, PhD, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- Hôpital Pitié-Salpêtriere, Paris, France

REFERENCES:
- [Background] Sole-Lleonart C, Rouby JJ, Chastre J, Poulakou G, Palmer LB, Blot S, Felton T, Bassetti M, Luyt CE, Pereira JM, Riera J, Welte T, Roberts JA, Rello J. Intratracheal Administration of Antimicrobial Agents in Mechanically Ventilated Adults: An International Survey on Delivery Practices and Safety. Respir Care. 2016 Aug;61(8):1008-14. doi: 10.4187/respcare.04519. Epub 2016 Mar 8. PMID 26957647
- [Background] Sole-Lleonart C, Rouby JJ, Blot S, Poulakou G, Chastre J, Palmer LB, Bassetti M, Luyt CE, Pereira JM, Riera J, Felton T, Dhanani J, Welte T, Garcia-Alamino JM, Roberts JA, Rello J. Nebulization of Antiinfective Agents in Invasively Mechanically Ventilated Adults: A Systematic Review and Meta-analysis. Anesthesiology. 2017 May;126(5):890-908. doi: 10.1097/ALN.0000000000001570. PMID 28248714
- [Background] Rello J, Rouby JJ, Sole-Lleonart C, Chastre J, Blot S, Luyt CE, Riera J, Vos MC, Monsel A, Dhanani J, Roberts JA. Key considerations on nebulization of antimicrobial agents to mechanically ventilated patients. Clin Microbiol Infect. 2017 Sep;23(9):640-646. doi: 10.1016/j.cmi.2017.03.018. Epub 2017 Mar 25. PMID 28347790
- [Background] Sole-Lleonart C, Roberts JA, Chastre J, Poulakou G, Palmer LB, Blot S, Felton T, Bassetti M, Luyt CE, Pereira JM, Riera J, Welte T, Qiu H, Rouby JJ, Rello J; ESGCIP Investigators. Global survey on nebulization of antimicrobial agents in mechanically ventilated patients: a call for international guidelines. Clin Microbiol Infect. 2016 Apr;22(4):359-364. doi: 10.1016/j.cmi.2015.12.016. Epub 2015 Dec 23. PMID 26723563